CLINICAL TRIAL: NCT01505244
Title: Before-School Physical Activity Intervention in Elementary School Children: A Pilot Study
Brief Title: Before-School Physical Activity Intervention in Elementary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Connie Tompkins, PhD, Assistant Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M12-031
Record Dates: First submitted 2011-12-27; First posted 2012-01-06 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Activity (Experimental): Before-school moderate to vigorous physical activity 3 days/week
  Interventions: Behavioral: Before-School Physical Activity

INTERVENTIONS:
Behavioral: Before-School Physical Activity — 3 days/week of before-school moderate to vigorous physical activity

SUMMARY:
Children in the U.S. exhibit low levels of physical activity. In addition to the overall physical health and fitness benefits with increasing levels of physical activity, improvements in academic performance, mental cognition, and behavior may occur. Despite these benefits, opportunities for children to participate in physical activity are being reduced, particularly in schools.

The proposed study is a pilot program with approximately 100 children ages 7-11 years expected to participate. All study participants will partake in a testing and measures session which will include body composition measures, nutrition and physical activity questionnaires, and curriculum-based measures. Following the first testing and measures session, 50 of the 100 children will participate in a 10-12 week, before-school, moderate to vigorous physical activity (MVPA) program. This program will consist of non-competitive, MVPA and occur 3 days/week at their school. Subsequent to the physical activity program, all 100 children will then participate in a follow-up testing and measures session.

The objective of this proposed pilot study is to determine the feasibility of implementing a before-school, physical activity program as well as explore the effect the program may have on academic performance and health measures.

DETAILED DESCRIPTION:
The current guidelines for physical activity recommend that children should partake in regular, moderate to vigorous intensity physical activity for 60 minutes or more each day. Unfortunately, children in the U.S. are not meeting these goals. Moreover, physical inactivity in these children is considered a significant, contributing factor to childhood overweight and obesity. In addition to the importance of physical activity for overall physical health and fitness, classroom behavior, academic skills, and attention may also improve in children with increasing physical activity. There appears to be a positive association between physical activity and academic performance, mental cognition, and behavior in children, however, further research to delineate the ideal duration and intensity is warranted particularly in elementary school children. As schools in recent years have eliminated recess and/or physical education due to growing pressure to increase academic scores, creative solutions to engage children in physical activity are desperately needed. And with the vast majority of children's time spent in school, this may be the ideal location for implementing physical activity interventions.

The purpose of this pilot study is to determine the feasibility of implementing a before-school, physical activity program. Furthermore, the effect the physical activity program may have on academic performance, and health measures will also be examined through several methods.

The results of the proposed study may help design future physical activity interventions and provide insight to the relationship between physical activity and academic performance.

ELIGIBILITY:
Inclusion Criteria:

* 3rd, 4th, or 5th grader currently attending Malletts Bay school
* Group A participants only: Approval to participate in a moderate to vigorous physical activity program from the child's pediatrician

Exclusion Criteria:

* Children will only be excluded from the study if both groups have reached their maximum capacity (n=50 in each group).
* Group A participants only: Approval to participate in a moderate to vigorous physical activity program not received from the child's pediatrician
* If a child has a known handicap and/or other medical condition and requires individualized education program (IEP) assistance, then the child may be excluded from the study if IEP accommodations are not available.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in curriculum-based measures at 12 weeks | 12 weeks
  The curriculum-based measures are unique methods of academic performance as these are sensitive to and are validated to monitor progress. Curriculum-based measures are easy to administer, can be given as often as wanted/needed, and provide immediate feedback. Progress monitoring focuses on individualized decision making in general and special education with respect to academic skill development at the elementary grades. Progress monitoring can be conducted frequently and is designed to estimate rates of improvement.

SECONDARY OUTCOMES:
Change from baseline in health-related measures at 12 weeks | 12 weeks
  Health-related measures will be measured at baseline as well as 12 weeks to assess changes in weight (kg), height (cm), waist, hip, and neck circumferences (cm), resting heart rate (bpm), and blood pressure (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Connie L Tompkins, PhD, Principal Investigator — University of Vermont
Locations (1):
- Malletts Bay School, Colchester, Vermont, United States

REFERENCES:
- [Derived] Tompkins CL, Hopkins J, Goddard L, Brock DW. The effect of an unstructured, moderate to vigorous, before-school physical activity program in elementary school children on academics, behavior, and health. BMC Public Health. 2012 Jul 5;12:300. doi: 10.1186/1471-2458-12-300. PMID 22537028